CLINICAL TRIAL: NCT01294917
Title: Comparison of a New AMO MPS to Existing Contact Lens Regimens
Brief Title: Comparison of a New Abbott Medical Optics (AMO) Multi-Purpose Solution (MPS) to Existing Contact Lens Regimens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Optics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: COBR-305-9608
Record Dates: First submitted 2011-02-10; First posted 2011-02-14 (Estimated); Results first posted 2012-05-14 (Estimated); Last update posted 2017-03-06 (Actual); Status verified 2017-01

CONDITIONS: Normal Contact Lens Wearers

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Investigational MPS (Experimental): AMO Investigational MPS.
  Interventions: Device: Multi-purpose disinfecting solution
- Clear Care (Active Comparator): Peroxide-based lens care regimen.
  Interventions: Device: Clear Care
- Opti-Free RepleniSH (Active Comparator): Multi-purpose disinfecting solution (Alcon).
  Interventions: Device: Opti-Free RepleniSH

INTERVENTIONS:
Device: Multi-purpose disinfecting solution — For the cleaning, rinsing, and storage of soft contact lenses.
  Arms: Investigational MPS
Device: Clear Care — Peroxide-based regimen for cleaning and disinfecting soft contact lenses.
  Arms: Clear Care
Device: Opti-Free RepleniSH — Multi-purpose disinfecting solution for the cleaning, rinsing and storing of soft contact lenses.
  Arms: Opti-Free RepleniSH

SUMMARY:
Crossover clinical evaluation three contact lens care regimens used for one month with Acuvue Oasys lenses.

DETAILED DESCRIPTION:
This is a three-arm crossover clinical evaluation of 40 subjects who will use each of three contact lens care regimens for one month with Acuvue Oasys lenses. The subjects will be randomized on the order of solutions used: Investigational MPS, ClearCare, and Opti-Free RepleniSH MPS.

ELIGIBILITY:
Inclusion Criteria:

* Is at least 17 years of age and has full legal capacity to volunteer;
* Has read and signed an information consent letter;
* Is willing and able to follow instructions and maintain the appointment schedule;
* Has had an ocular examination in the last two years;
* Is a current soft lens wearer using either two-week or monthly replacement lenses;
* Is correctable to a visual acuity of 6/7.5 (20/25) or better (both eyes) with their habitual vision correction (either spectacles or contact lenses);
* Has normal binocular vision (no strabismus, no amblyopia);
* Has clear corneas and no active ocular disease;
* Has a distance contact lens prescription between +8.00 diopters (D) to -12.00 D and a successful fit with the study lenses;
* Has astigmatism less than or equal to -1.00 D;
* Agrees to wear the study lenses on a daily wear basis.

Exclusion Criteria:

* Has any active ocular disease;
* Has any clinically significant lid, conjunctival, or corneal abnormalities that may affect a study outcome variable;
* Has undergone corneal refractive surgery;
* Has a systemic condition that may affect a study outcome variable;
* Is using any systemic or topical medications that may affect ocular health;
* Has known sensitivity to the diagnostic pharmaceuticals to be used in the study;
* Is pregnant or lactating;
* Is participating in any other clinical or research study that may affect a study outcome variable;
* Currently wears daily disposable lenses or extended wear lenses.

Min Age: 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-02; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Craig Woods, MOptom, Principal Investigator — University of Waterloo
Locations (1):
- Centre for Contact Lens Research, Waterloo, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Groups:
- All Participants: All subjects received each of 3 study solutions for one month each for the daily care of their soft contact lenses. Subjects were randomized to six possible sequences of use of each study solution: AMO Investigational MPS, Clear Care and OptiFree ReplenisH MPS.
Period: Overall Study
Arm/Group | All Participants
Started | 42
Received Investigational MPS | 36
Received Clear Care | 36
Received OptiFree RepleniSH MPS | 36
Completed | 36
Not Completed | 6
Not completed — Relocation | 5
Not completed — Inconvenience | 1

BASELINE CHARACTERISTICS:
Arm/Group | All Participants
Number analyzed (Participants) | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 41
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.1 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33
  Male | 9
Region of Enrollment [Number; unit: participants]
  Canada | 42

OUTCOME MEASURES:

1. Primary Outcome: Corneal Staining
Description: Corneal staining will be assessed with sodium fluorescein dye on the ocular surface. The cornea is split into 5 sections, each section is evaluated by staining type, depth, and extent is graded on a 0 to 100 scale with higher scores indicating more staining. The possible total range for the total score per eye is 0 to 50,000 (100x100x100=10,000 per section) with values higher than 1200 being clinically relevant.
Time Frame: 4 weeks
Population: Only subjects that completed all three arms were included in analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- AMO Investigational MPS: All subjects received the AMO Investigational MPS for one month for the care of their soft contact lenses.
- Clear Care: All subjects received the Clear Care for one month for the care of their soft contact lenses.
- OptiFree RepleniSH MPS: All subjects received the OptiFree RepleniSH MPS for one month for the care of their soft contact lenses.
Arm/Group | AMO Investigational MPS | Clear Care | OptiFree RepleniSH MPS
Number analyzed (Participants) | 36 | 36 | 36
units on a scale | 184 (381.6) | 46.6 (91.3) | 77.8 (131.7)

2. Secondary Outcome: Subjective Lens Wearing Comfort
Description: This will be assessed by a questionnaire on patient-perceived lens comfort and any symptoms of discomfort on a 0 to 100 scale.
Time Frame: 4 weeks
Reporting Status: Not Posted

3. Secondary Outcome: Dryness
Description: This will be assessed by the tear break-up time on the lens surface, measured in seconds.
Time Frame: 4 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | All Participants
Serious Adverse Events (participants affected / at risk) | 0/42
Other Adverse Events (participants affected / at risk) | 0/42

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No